CLINICAL TRIAL: NCT00415350
Title: Bronchiectasis and Long Term Azithromycin Treatment: A Randomised Placebo-controlled Trial Studying Disease Modifying Effects of Immunomodulating Treatment
Brief Title: Bronchiectasis and Long Term Azithromycin Treatment
Acronym: BAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: W.G.Boersma (Other)
Responsible Party: Sponsor-Investigator, W.G.Boersma, Doctor, MD, Medical Center Alkmaar
Organization: Medical Center Alkmaar (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2006-MCA1; BAT-2006
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Bronchiectasis; Inflammation
Keywords: Bronchiectasis; Macrolide; Azithromycin; Antibiotic prophylaxis; Immunomodulation; Inflammation; Lung function; Sputum; Bacterial colonization
MeSH Terms: conditions — Bronchiectasis; Inflammation | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin treatment 1 (Active Comparator)
  Interventions: Drug: Azithromycin
- Placebo 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin Tablet 250 mg daily
  Arms: Azithromycin treatment 1
Other: Placebo — Placebo tablet 1 daily
  Arms: Placebo 2

SUMMARY:
1. SUMMARY

Rationale: Patients with bronchiectasis often experience lower respiratory tract infections with progression of symptoms and decline in quality of life. Macrolides, as has been shown in panbronchiolitis and cystic fibrosis, may break or weaken the link between infection and inflammation resulting in an improvement of symptoms. Also the number of exacerbations may lowered.

Objective: A reduction in number of infective exacerbations and improvement in lung function by AZT treatment are the primary objectives. Secondary objectives that will be evaluated are: symptoms score, quality of life, inflammatory parameters, bacterial colonisation, and adverse events.

Study design: Randomised double blind multicenter study in the Netherlands. Patients will be stratified for colonisation with P.aeruginosa.

Study population: Patients with bronchiectasis demonstrated by high-resolution computed tomography (HR-CT) scan or bronchography.

Intervention: Patients receive Azithromycin 250mg(p.o.) once daily or placebo.

Main study parameters/endpoints: Reduction in number exacerbations, defined as increase symptoms such as dyspnoea, coughing, and sputum production for which a course of prednisolone and/or antibiotic is needed. Change in lung function parameters (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC]) measured by spirometry is the other primary endpoint.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk of participating in this study is low. Laboratory, radiographic examinations, and pulmonary function tests are commonly used as diagnostic procedures during outpatients visits and during exacerbations. Adverse effects in maintenance treatment with AZT are usually mild and mainly gastrointestinal. Sometimes rash and abnormal liver function tests are observed. A better quality of life will probably be the beneficial effect of long term treatment with AZT. This will be achieved by a reduction in respiratory and non-respiratory symptoms and number of exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 ≥ years
* Bronchiectasis diagnosed by plain bronchography or high resolution computer tomography.
* Minimal 3 lower respiratory tract infections (LRTI) treated with oral/intravenous (IV) antibiotics in the year preceding the study inclusion.
* The presence of chronic respiratory symptoms such as cough, dyspnoea, expectoration of sputum.
* At least one positive sputum culture in the preceding year.
* Informed consent

Exclusion Criteria:

* Previous ( ≥ 4 weeks) prolonged macrolide therapy.
* Pregnant or lactating women.
* Allergy to macrolides.
* Intolerance to macrolides.
* Liver disease (alanine transaminase and/or aspartate transaminase levels 2 or more times the upper limit of normal).
* Use of antibiotics within 14 days of screening.
* Use of oral or IV corticosteroids (≥ 30 mg prednisolone/daily) within 30 days of screening.
* Other research medication started 2 months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Does prolonged antibiotic treatment with AZM reduce the number of bacterial exacerbations in patients with bronchiectasis? | 1 year
Does treatment with AZM increase lung function parameters (Δ FEV1, Δ FVC )? | 1 year

SECONDARY OUTCOMES:
Is there any improvement in symptom score during treatment with AZM? | 1 year
What is the effect of AZM on bacterial colonisation? | 1 year
Does treatment with AZM reduce inflammatory parameters? | 1 year
Does treatment with AZM change the quality of life? | 1 year
Is there any differences in adverse events between AZM and placebo treatment? | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: W.G. Boersma, MD,PHD, Study Director — Medical Center Alkmaar, dep. Pulmomary Diseases
Locations (16):
- Netherlands (16):
  - Alkmaar Medical Center, Alkmaar, N-H
  - AMC, Amsterdam
  - St Lucas Andreas Ziekenhuis, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Deventer Ziekenhuis, Deventer
  - U.L.C. Dekkerswald, Groesbeek
  - University Hospital Groningen (UMCG), Groningen
  - Atrium Medisch Centrum, Heerlen
  - Tergooi Ziekenhuizen, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - MC Leeuwarden, Leeuwarden
  - Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Diakonessenhuis, Utrecht
  - Viecuri MC, Venlo
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Terpstra LC, Altenburg J, Mohamed Hoesein FA, Bronsveld I, Go S, van Rijn PAC, De Jong PA, Heijerman HGM, Boersma WG. The effect of maintenance azithromycin on radiological features in patients with bronchiectasis - Analysis from the BAT randomized controlled trial. Respir Med. 2022 Feb;192:106718. doi: 10.1016/j.rmed.2021.106718. Epub 2021 Dec 28. PMID 34974413
- [Derived] Altenburg J, de Graaff CS, Stienstra Y, Sloos JH, van Haren EH, Koppers RJ, van der Werf TS, Boersma WG. Effect of azithromycin maintenance treatment on infectious exacerbations among patients with non-cystic fibrosis bronchiectasis: the BAT randomized controlled trial. JAMA. 2013 Mar 27;309(12):1251-9. doi: 10.1001/jama.2013.1937. PMID 23532241